CLINICAL TRIAL: NCT00033969
Title: Complex Regional Pain Syndrome Proteomics Study
Brief Title: Study of Proteins Associated With Complex Regional Pain Syndrome
Status: Terminated | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020169; 02-NR-0169
Record Dates: First submitted 2002-04-17; First posted 2002-04-18 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-10-23

CONDITIONS: Complex Regional Pain Syndromes; Healthy
Keywords: CRPS; RSD; Causalgia; Chronic Pain; Neuropathic Pain; Normal Control; Complex Regional Pain Syndrome; Healthy Volunteer; HV
MeSH Terms: conditions — Complex Regional Pain Syndromes; Causalgia; Chronic Pain; Neuralgia

SUMMARY:
This study will try to learn more about complex regional pain syndrome, or CRPS (previously known as reflex sympathetic dystrophy, spreading neuralgia, and sympathalgia), by examining the release of small proteins in the blood of patients with this condition. Patients with CRPS usually have three types of symptoms:

* Sensory abnormalities increased sensitivity to pain or a painful reaction to a harmless stimulus
* Perfusion abnormalities alterations in blood flow, temperature abnormality, swelling, decrease or increased nail growth, and hair and skin changes
* Motor abnormalities weakness, guarding (Holding the limb in such a fashion that it minimizes accidental or intentional contact from possible sources of pain), and atrophy (wasting)

The cause of CRPS is unknown, and there are no definitive diagnostic tests for the condition. Because early treatment improves the prognosis of CRPS, a test that enables early diagnosis would be important for optimal medical management. The findings of this study may contribute to the development of such a test and possibly new drug treatments.

Normal healthy volunteers and patients of any age with complex regional pain syndrome who are in otherwise good general health may be eligible for this study.

Participants will have a medical history, physical examination and collection of a blood sample. They will fill out several questionnaires, providing information on their health, personality, mood, pain levels, and symptoms. Participation in the study requires one outpatient clinic visit.

DETAILED DESCRIPTION:
The etiology of Complex Regional Pain Syndrome (CRPS) is unknown but a patient typically presents with a triad of clinical findings: sensory abnormalities, perfusion abnormalities and alterations in motor function. Since some of these findings are seen in the other disease states, the diagnosis is often not clear. A response to a sympathetic ganglion block (stellate or lumbar) is also suggestive of the disorder. However, there is no definitive diagnostic test for CRPS. Experience has shown that early aggressive treatment improves the prognosis. Therefore, tests that facilitate the early diagnosis would have important clinical implications.

Advances in laboratory techniques allow analysis of clinical samples to identify protein or patterns of protein changes associated with a disease state. Patients suffering with CRPS who are currently seen in a pain clinic will be asked to participate in this study. The subjects will complete a brief symptom survey, be examined by a co-investigator to document sensory, temperature and trophic changes, and have a blood sample collected for protein and gene expression (RNA) analysis. Blood samples from age-matched controls will be collected from non-CRPS patients. Fifty patient samples collected from each group will be analyzed and used to teach the diagnostic software and an additional 20 samples (10 controls, 10 CRPS patients) will be used to validate diagnostic accuracy.

ELIGIBILITY:
* INCLUSION CRITERIA
* Male or female patients referred by their physician with the diagnosis of CRPS criteria as outlined by Stanton-Hicks et al.

OR

* Healthy volunteers will be screened according to the eligibility criteria as specified in the appendix (see Healthy Subject Eligibility).
* Age restrictions: Patients and volunteers must be (Bullet)18 years of age at the time of enrollment. There is no upper limit for age of inclusion.
* Good general health (other disease states could may confound the results see exclusion criteria)
* Willing to have blood drawn
* Willing to have behavioral measures
* Willing to provide a directed medical history
* There is expected to be a greater number of females than males being recruited to this study since there is a much higher occurrence of CRPS in women. Additionally, it is expected to be equal across all ethnic groups. However, we do not anticipate requiring any special recruiting strategies for specific gender or ethnic groups.

EXCLUSION CRITERIA

* Contraindication to blood screening
* Advanced disease other than the CRPS (cardiovascular, liver, kidney disease ASA III or above excluding CRPS) that may cause a theoretical inclusion of samples resulting in confounding results.
* Pregnant and lactating women.

No exclusions will be made based on race, gender, or religion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2002-04-15; Study Completion 2014-10-23

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Mannes, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bichsel VE, Liotta LA, Petricoin EF 3rd. Cancer proteomics: from biomarker discovery to signal pathway profiling. Cancer J. 2001 Jan-Feb;7(1):69-78. PMID 11269650
- [Background] Bittner M, Meltzer P, Chen Y, Jiang Y, Seftor E, Hendrix M, Radmacher M, Simon R, Yakhini Z, Ben-Dor A, Sampas N, Dougherty E, Wang E, Marincola F, Gooden C, Lueders J, Glatfelter A, Pollock P, Carpten J, Gillanders E, Leja D, Dietrich K, Beaudry C, Berens M, Alberts D, Sondak V. Molecular classification of cutaneous malignant melanoma by gene expression profiling. Nature. 2000 Aug 3;406(6795):536-40. doi: 10.1038/35020115. PMID 10952317
- [Background] Chelimsky TC, Low PA, Naessens JM, Wilson PR, Amadio PC, O'Brien PC. Value of autonomic testing in reflex sympathetic dystrophy. Mayo Clin Proc. 1995 Nov;70(11):1029-40. doi: 10.4065/70.11.1029. PMID 7475332